CLINICAL TRIAL: NCT01999374
Title: Long Term Follow up of Recipients of Functional Islet Allografts
Status: Recruiting | Type: Observational
Sponsor: Rodolfo Alejandro (Other)
Responsible Party: Sponsor-Investigator, Rodolfo Alejandro, Professor of Medicine, University of Miami
Organization: University of Miami (Other)
Other Study IDs: 20130034
Record Dates: First submitted 2013-11-25; First posted 2013-12-03 (Estimated); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Since its inception, the Diabetes Research Institute (DRI) has made significant contributions to the field of diabetes, pioneering many of the techniques used in diabetes centers around the world. Through several clinical trials, DRI has demonstrated that diabetes can be successfully reversed as a result of islet cell transplant.

Over the years the following protocols in islet cell transplantation have been initiated: 2000/0329; 2000/0196; 2004/0205; 2000/024; 2006/0200; 2006/0508; 2006/0210.

All of the studies listed above will be source of study subjects for this study. Approximately 30 subjects are expected to be enrolled and followed in this trial.

After islet-cell transplantation in the parent studies, each subject receives maintenance immunosuppressive medications.

The purpose of this protocol is to collect additional follow-up for safety and efficacy from subjects with graft function after their completion in their parent study. It is expected that most subjects will retain measurable islet function and, in the islet-alone studies, continue to receive immunosuppressive medications at the time of completing their parent study.

DETAILED DESCRIPTION:
To provide long term follow up in subjects with functional islet allografts.

ELIGIBILITY:
Inclusion Criteria:

1. Participation in any of the following parent studies: 2000/0329; 2000/0196; 2004/0205; 2000/0024; 2006/0200; 2006/0508; 2006/0210
2. A functioning pancreatic islet graft (absence of graft failure as defined in parent study) requiring immunosuppression.
3. Willingness of participants to continue to use an approved method of contraception during and 4 months after study participation.
4. Ability to provide written informed consent.

Exclusion Criteria:

1. For female subjects: Positive pregnancy test, presently breast-feeding, or unwillingness to use effective contraceptive measures for the duration of the study and 4 months after discontinuation. For male subjects: intent to procreate during the duration of the study or within 4 months after discontinuation or unwillingness to use effective measures of contraception. Oral contraceptives, Norplant®, Depo-Provera®, and barrier devices with spermicide are acceptable contraceptive methods; condoms used alone are not acceptable.
2. Any medical condition that, in the opinion of the investigator, will interfere with safe participation in the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject with Type 1 diabetes mellitos status post islet transplantation
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2013-03; Primary Completion 2027-03 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Duration of sustained islet allograft function | 3 years
  The primary endpoint is duration of sustained islet allograft function as determined by evidence from Mixed Meal Tolerance Test of c-peptide production. A c-peptide level >=0.3 ng/ml at 0, 60, or 90 minutes will be considered evidence of islet allograft function.

CONTACTS AND LOCATIONS:
Overall Officials: Rodolfo Alejandro, MD, Principal Investigator — University of Miami
Locations (1):
- Diabetes Research Institute, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rios P, Baidal D, Lemos J, Camhi SS, Infante M, Padilla N, Alvarez Gil AM, Fuenmayor V, Ambut J, Qasmi FA, Mantero AM, Cayetano SM, Ruiz P, Ricordi C, Alejandro R. Long-term Persistence of Allosensitization After Islet Allograft Failure. Transplantation. 2021 Nov 1;105(11):2490-2498. doi: 10.1097/TP.0000000000003635. PMID 33481552